CLINICAL TRIAL: NCT00289809
Title: A Perspective Phase I and II Trial of Liposome-encapsulated Doxorubicin (TLC D-99) in Combination With Ifosfamide in Patients With Metastatic Soft Tissue Sarcoma
Brief Title: TLC D-99 and Ifosfamide in Metastatic Soft Tissue Sarcoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Dr. Armando Santoro, Istituto Clinico Humanitas
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2005-001; EUDRACT 2005-004569-40
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2009-12

CONDITIONS: Sarcoma, Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: combination of TLC D-99 and Ifosfamide — * TLC D-99: 40 mg/m2 Day 1 every 3 weeks;
  * Ifosfamide: 3000 mg/m2 Day 1, 2, 3 every 3 weeks

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of the TLC D-99 combined with ifosfamide and then the efficacy of this combination in terms of overall response rate, time to progression and time of response

DETAILED DESCRIPTION:
The Maximum Tolerated Dose of the combination was determined and the Phase I terminated.

Then, Phase II study started.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of soft tissue sarcoma metastatic or recurrent after 6 months from the last chemotherapy
* Age >/=18 yrs
* PS </=2
* Disease detectable almost for 1 dimension
* Life expectancy >/=3 mos
* Minimum 4 wks from last radiotherapy
* Adequate medullary, liver, and renal functions
* Normal LVEF
* Written Informed Consent

Exclusion Criteria:

* Pregnant or breast-feeding patients
* Serious concomitant disease or not controlled infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose (MTD) of combination of TLC D-99 and Ifosfamide | Definition of TDL
Phase II: Response rate (CR/PR or SD) | Tumor assessment

SECONDARY OUTCOMES:
Phase II: time to progression, duration of response, overall survival | Tumor assessment, follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy